CLINICAL TRIAL: NCT03704779
Title: Effectiveness of a Multimodal Mindfulness Program to Alleviate Graduate Student Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Sharon Gutman, Professor of Rehabilitation and Regenerative Medicine (OT, Rehab & Regenerative Med), Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAAS0303
Record Dates: First submitted 2018-10-10; First posted 2018-10-15 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Stress
Keywords: Mindfulness; Student

STUDY DESIGN:
Intervention Model Description: Intervention will be implemented over 8 consecutive weeks and will consist of experiential mindfulness activities that can be accessed in-person and online. In-person mindfulness activities will be available twice per week and last approximately 40 minutes in length. Mindfulness meditation videos posted online will be available 24/7 and last 10-45 minutes. Students will be asked to participate in one 40-minute in-person and four 10-minute online mindfulness activities per week (total of 1 hour and 20 minutes per week).
  Week 1. Progressive muscle relaxation, mindfulness meditation, guided imagery.
  Week 2. Mindfulness: Zen garden, painting, craftwork.
  Week 3. Active Meditation: yoga, Tai Chi.
  Week 4. Aromatherapy.
  Week 5. Addiction Information and Management Strategies.
  Week 6. Positive Psychology Strategies: cognitive reframing techniques.
  Week 7. Self-Compassion Strategies: walking meditation, nutritious snacks, self-massage.
  Week 8. Pet Therapy.
Who Masked: Outcomes Assessor
Masking Description: Data collectors will be masked to participant group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multimodal Mindfulness Activity Program (Experimental): Students assigned to the intervention will receive 8 weeks of the mindfulness activity intervention.
  Interventions: Behavioral: Multimodal mindfulness activity program
- Control Group (No Intervention): Students assigned to the control group will not receive any intervention.

INTERVENTIONS:
Behavioral: Multimodal mindfulness activity program — This program will provide the opportunity for participants to engage in in-person and online activities. The in-person activities will be held from 12:00 pm to 12:45 pm in the Georgian Physical Therapy Lab (and offered twice per week). The online activities will be available at all times during the study at convenience. There are one 40-minute in-person and four 10-minute online mindfulness activities per week (combined time of 1 hour and 20 minutes per week).
  In-person activities will consist of mindfulness activities including guided imagery meditation, yoga, Tai Chi, progressive muscle relaxation, creating a Zen garden, aromatherapy, journaling, self-massage, and pet therapy. Online materials will additionally include guided and unguided meditations.
  Arms: Multimodal Mindfulness Activity Program

SUMMARY:
The purpose of this pilot study is to develop and assess a multimodal mindfulness activity program for physical and occupational therapy students intended to teach management of stressors impacting educational performance. This study will use a two group, randomized controlled design in which approximately 25 students will be randomized to an intervention group and 25 to a control group. Intervention will be implemented in an 8-week period with pre- and post-study measures administered at 1-week prior to and 1-week following intervention.

DETAILED DESCRIPTION:
College students have reported increasing stress levels in the last 5 years with 1 in 6 students experiencing anxiety levels that adversely impact school function. This study's intervention uses a variety of media and both online and in-person delivery strategies. For example, students will have the opportunity to participate in yoga, Tai Chi, guided imagery meditation, creative arts, journaling, and pet therapy. Students will additionally have the opportunity to participate in activities delivered through online media and accessible at all times throughout the study. Approximately 50 occupational and physical therapy students will be recruited to participate in this study. Half will be selected by chance to participate in the 8-week program; the remaining half will be selected by chance to participate in a non-intervention group in which they do not receive the program but are still assessed at pre- and post-program to measure perceived stress levels. It is anticipated that study results will provide information to educational institutions to help students better manage stress levels.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be student volunteers in the Columbia University Physical and Occupational Therapy Programs.
* Students must be in their first or second year, second semester in order to compare GPA pre- and post-intervention.

Exclusion Criteria:

* Students who are practiced meditators or who have prior experience with mindfulness training will be excluded from study participation, as such previous experience could bias intervention results.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-04-11 (Actual); Study Completion 2019-04-11 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale | 10 minutes
  The Perceived Stress Scale (PSS) is a 10-item, 5-point, self-report Likert scale (0 = no stress, 5 = high stress) that requires 5 minutes to complete. The scale yields a total score ranging from 0 (no stress) to 50 (highest stress) with scores 25+ indicating a possible stress disorder. The PSS measures stress level in the last month and was intended for use by community-dwelling adults.

SECONDARY OUTCOMES:
Student Stress Management Questionnaire | 10 minutes
  The Student Stress Management Questionnaire (SSMQ) is a 12-item, 5-point Likert scale (0 = no stress, 5 = high stress) that requires 5 minutes to complete. The scale yields a total score ranging from 0 (no stress) to 60 (highest stress) with scores 40+ indicating a possible stress disorder. The SSMQ measures stress level in the last month and was intended for use by college students.
Daily Log | 10 minutes
  The daily log is a 6-item questionnaire that allows students to record the number and length of mindfulness activities in which they participated that day. Students also report their level of stress before and after participation using a 5-point Likert scale (0 = no stress, 5 = high stress). Scores of 15+ indicate higher stress levels.
Grade Point Average (GPA) | 5 minutes
  GPA will be calculated for the semester prior to and directly after study participation.
Number of Student Wellness Center Visits | 5 minutes
  The number of Student Wellness Center visits prior to and directly after study participation will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon A Gutman, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No